CLINICAL TRIAL: NCT04742179
Title: Fighting Climate Change: Urban Greennes, Active Mobility and Health Co-benefits.
Acronym: CLIMACTIONS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Research Manager, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11/2020
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Respiratory and Allergic Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The children belonging to the classes of the school complex undergoing the maintenance intervention.
  Interventions: Other: Manteinance and care intervention on the green areas.
- Control group (No Intervention): The children belonging to the classes of the school complex that will not undergo the maintenance intervention.

INTERVENTIONS:
Other: Manteinance and care intervention on the green areas. — Manteinance and care intervention on the green areas.
  Arms: Experimental group

SUMMARY:
This is a prospective, non-randomized, controlled, interventional study aiming to assess, in a primary school in the city of Palermo, the health effects of a maintenance and care intervention of the school's green areas.

All children of the third, fourth and fifth classes of two school complexes of the same primary school will be selected. One complex will undergo maintenance and care of the green areas and gardens inside the school. The other complex will serve as a control group and will not undergo any intervention.

The study will involve three phases.

1. During the first phase (prior to the intervention) respiratory and allergic symptoms will be assessed through a standardized questionnaire to be administered to students, parents and teachers in both the school complexes.
2. During the second phase, the maintenance and care intervention plan will be implemented in the experimental complex.
3. During the third phase, 1 week after the maintenance intervention, respiratory and allergic symptoms will be re-assessed through a standardized questionnaire to be administered to the same students, parents and teachers in both the school complexes.

ELIGIBILITY:
Inclusion Criteria:

* male or female gender
* age between 7 and 11 years

Exclusion Criteria:

* no exclusion criteria

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms at baseline | Before the maintenance intervention
  Presence of asthma symptoms before the maintenance intervention
Rhinitis symptoms at baseline | Before the maintenance intervention
  Presence of rhinitis symptoms before the maintenance intervention
Conjunctivitis symptoms at baseline | Before the maintenance intervention
  Presence of conjunctivitis symptoms before the maintenance intervention
Asthma symptoms at follow-up | 7 days after the maintenance intervention
  Presence of asthma symptoms after the maintenance intervention
Rhinitis symptoms at follow-up | 7 days after the maintenance intervention
  Presence of rhinitis symptoms after the maintenance intervention
Conjunctivitis symptoms at follow-up | 7 days after the maintenance intervention
  Presence of conjunctivitis symptoms after the maintenance intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Translational Pharmacology, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No